CLINICAL TRIAL: NCT01958307
Title: Healthy Living in Pregnancy
Acronym: GeliS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GEL-1309--2500-S
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Lifestyle; Weight Gain; Pregnancy
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Lifestyle intervention
  Interventions: Behavioral: Lifestyle intervention
- No intervention (No Intervention): Standard prenatal care, short information leaflet about healthy lifestyle in pregnancy

INTERVENTIONS:
Behavioral: Lifestyle intervention — The intervention program consists of four individual counseling modules focusing on diet, physical activity and weight monitoring (12th-16th, 16th-20th, 30th-34th week of gestation and 6th-8th week postpartum). The counseling sessions are given by carefully trained midwives or medical staff in combination with prenatal visits and follow a standardized curriculum. Women are provided with brochures including a list of adequate prenatal exercise programs and a pedometer. Furthermore, they receive a chart personalized according to their baseline BMI category to monitor weight development.
  Arms: Intervention

SUMMARY:
Multicenter and multidisciplinary public health project in 10 regions of Bavaria, a federal state of Germany, targeting maternal and fetal health. The objective of this trial is to evaluate the efficacy of a lifestyle intervention program focusing on diet, physical activity and weight monitoring during pregnancy. The intervention comprises 4 individual counseling sessions addressing healthy living. Primary outcome: gestational weight gain. Secondary outcomes are pregnancy and obstetric complications like gestational diabetes and rate of caesarean sections as well as offspring health.

The lifestyle intervention program is adapted to the German health care system to allow an immediate implementation after successful evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 12th week of gestation
* Age: 18 years to 43 years
* Prepregnancy BMI ≥ 18.5 kg/m2 and ≤ 40.0 kg/m2
* Sufficient German language skills
* Written informed consent

Exclusion Criteria:

* Multiple pregnancy
* Any condition preventing physical activity such as placenta praevia, persistent bleeding, cervical incompetence
* Prepregnancy diabetes or early diagnosed gestational diabetes
* Uncontrolled chronic diseases (e.g. thyroid dysfunction)
* Psychiatric or psychosomatic diseases
* Any condition that may interfere with the study protocol

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2286 (Actual)
Dates: Start 2013-09; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 4 years
  Proportion of pregnant women showing excessive gestational weight gain according to Institute of Medicine (IOM) guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hauner, Prof. Dr., Principal Investigator — Else Kröner-Fresenius-Zentrum für Ernährungsmedizin
Locations (5):
- Germany (5):
  - AELF, Fachzentrum L 3.10 Ernährung/Gemeinschaftsverpflegung, Bayreuth
  - AELF, Fachzentrum L 3.10 Ernährung/Gemeinschaftsverpflegung, Fürstenfeldbruck
  - AELF, Fachzentrum L 3.10 Ernährung/Gemeinschaftsverpflegung, Fürth
  - AELF, Fachzentrum L 3.10 Ernährung/Gemeinschaftsverpflegung, Regensburg
  - AELF, Fachzentrum L 3.10 Ernährung/Gemeinschaftsverpflegung, Würzburg

REFERENCES:
- [Background] Rauh K, Gabriel E, Kerschbaum E, Schuster T, von Kries R, Amann-Gassner U, Hauner H. Safety and efficacy of a lifestyle intervention for pregnant women to prevent excessive maternal weight gain: a cluster-randomized controlled trial. BMC Pregnancy Childbirth. 2013 Jul 16;13:151. doi: 10.1186/1471-2393-13-151. PMID 23865624
- [Derived] Geyer K, Raab R, Hoffmann J, Hauner H. Development and validation of a screening questionnaire for early identification of pregnant women at risk for excessive gestational weight gain. BMC Pregnancy Childbirth. 2023 Apr 13;23(1):249. doi: 10.1186/s12884-023-05569-7. PMID 37055730
- [Derived] Raab R, Hoffmann J, Spies M, Geyer K, Meyer D, Gunther J, Hauner H. Are pre- and early pregnancy lifestyle factors associated with the risk of preterm birth? A secondary cohort analysis of the cluster-randomised GeliS trial. BMC Pregnancy Childbirth. 2022 Mar 21;22(1):230. doi: 10.1186/s12884-022-04513-5. PMID 35313852
- [Derived] Johar H, Hoffmann J, Gunther J, Atasoy S, Stecher L, Spies M, Hauner H, Ladwig KH. Evaluation of antenatal risk factors for postpartum depression: a secondary cohort analysis of the cluster-randomised GeliS trial. BMC Med. 2020 Jul 24;18(1):227. doi: 10.1186/s12916-020-01679-7. PMID 32703266
- [Derived] Hoffmann J, Gunther J, Geyer K, Stecher L, Rauh K, Kunath J, Meyer D, Sitzberger C, Spies M, Rosenfeld E, Kick L, Oberhoffer R, Hauner H. Effects of a lifestyle intervention in routine care on prenatal physical activity - findings from the cluster-randomised GeliS trial. BMC Pregnancy Childbirth. 2019 Nov 11;19(1):414. doi: 10.1186/s12884-019-2553-7. PMID 31711430
- [Derived] Kunath J, Gunther J, Rauh K, Hoffmann J, Stecher L, Rosenfeld E, Kick L, Ulm K, Hauner H. Effects of a lifestyle intervention during pregnancy to prevent excessive gestational weight gain in routine care - the cluster-randomised GeliS trial. BMC Med. 2019 Jan 14;17(1):5. doi: 10.1186/s12916-018-1235-z. PMID 30636636
- [Derived] Rauh K, Kunath J, Rosenfeld E, Kick L, Ulm K, Hauner H. Healthy living in pregnancy: a cluster-randomized controlled trial to prevent excessive gestational weight gain - rationale and design of the GeliS study. BMC Pregnancy Childbirth. 2014 Mar 28;14:119. doi: 10.1186/1471-2393-14-119. PMID 24678761